CLINICAL TRIAL: NCT07274956
Title: Is Pelvic Pain Severity Correlated With Nerve Fiber Density Within DIE Nodules?
Brief Title: Nerve Fiber Density in DIE Nodules & Pelvic Pain
Acronym: DIENerveDens
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Baris KAYA, Associate Professor, Başakşehir Çam & Sakura City Hospital
Other Study IDs: 2025-214; The authors BK and SHA (Other: Basakehir Cam ve Sakura City Hospital)
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Deep Infiltrating Endometriosis, Pelvic Pain, Dysmenorrhea Dyspareunia
Keywords: Deep infiltrating endometriosis; Pelvic pain; Dysmenorrhea; Dyspareunia; Nerve fiber density; SOX10
MeSH Terms: conditions — Pelvic Pain; Dysmenorrhea; Dyspareunia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DIE Nodule Pathology Cohort: Women (18-55 years) with surgically confirmed deep infiltrating endometriosis (DIE) who underwent standard-of-care resection (e.g., nodule excision, nerve-sparing hysterectomy ± salpingo-oophorectomy, and/or segmental bowel surgery when indicated). This is an observational, retrospective cohort; no investigational intervention is administered. The exposure of interest is nodule-level nerve fiber density, quantified on archived FFPE blocks by histopathology and immunohistochemistry (e.g., SOX10). Clinical data (demographics, gynecologic history, prior treatments) and patient-reported pain scores (VAS for dysmenorrhea, dyspareunia, dyschezia, dysuria, chronic pelvic pain) are abstracted from records. Primary analyses assess the association between nerve fiber density and pelvic pain severity/localization; secondary analyses explore relationships with lesion site/depth and other clinicopathologic features.

SUMMARY:
Deep infiltrating endometriosis (DIE) is a highly symptomatic form of endometriosis linked to severe dysmenorrhea, dyspareunia, dyschezia, dysuria, and chronic pelvic pain. Histologic studies suggest abundant neural elements in DIE nodules, but the relationship between nodule-level nerve fiber density and patient-reported pelvic pain remains insufficiently defined. This retrospective, cross-sectional study with prospective pathology re-review evaluates whether nerve fiber density in surgically excised DIE nodules correlates with pain severity and location. Women aged 18-55 who underwent surgery for DIE after inadequate response to medical therapy are included. Clinical data (demographics, gynecologic history, prior treatments) and standardized pain scores (VAS for pain domains) are abstracted from records. Archived blocks are recut; sections are stained with H&E and immunolabeled (e.g., SOX-10) to quantify neural profiles and derive a nerve fiber density metric per nodule. Primary endpoint: association between nerve fiber density and pain intensity/localization. Secondary endpoints: relationships with lesion site/depth and other clinicopathologic variables; exploratory discrimination of severe-pain phenotypes. Statistics (χ²/Fisher, t/Mann-Whitney, Kaplan-Meier/Cox if applicable) use two-sided p<0.05. This minimal-risk study uses existing records and archived tissue only; findings may inform counseling, nerve-sparing surgical planning, and future biomarker-driven, response-adapted trials.

DETAILED DESCRIPTION:
Deep infiltrating endometriosis (DIE) is a highly symptomatic phenotype of endometriosis that invades retrocervical, parametrial, rectovaginal, bowel, and other pelvic structures, and is frequently associated with severe dysmenorrhea, dyspareunia, dyschezia, dysuria, and chronic pelvic pain. Emerging evidence suggests that DIE nodules harbor abundant nerve fibers and may show perineural involvement, yet the relationship between intranodular nerve fiber density and patient-reported pelvic pain has not been defined with sufficient clinical granularity.

This retrospective, cross-sectional study with prospective pathology re-review investigates whether nerve fiber density within surgically excised DIE nodules correlates with the intensity and localization of pelvic pain. Eligible participants are women (18-55 years) operated for DIE after inadequate response to medical therapy (e.g., nodule excision, nerve-sparing hysterectomy ± salpingo-oophorectomy, ovarian surgery, and/or bowel resection when indicated). Demographic characteristics, obstetric/gynecologic history, prior surgeries and medical treatments, and standardized pain assessments (visual analogue scale [VAS] scores for dysmenorrhea, dyspareunia, dyschezia, dysuria, and chronic pelvic pain) are abstracted from the hospital information system.

All resected specimens are routinely fixed in buffered formalin and processed for histopathology. For this study, archived blocks from endometriotic foci are recut (3-µm sections) and stained with hematoxylin-eosin and immunohistochemically labeled with SOX-10 to visualize neural elements. Under ×200 magnification, the number of SOX-10-positive neural profiles within endometriotic foci is quantified, and mean nerve fiber counts (per evaluated field/area) are calculated to derive a nerve fiber density metric for each nodule. The primary endpoint is the association between nodule-level nerve fiber density and pain severity/localization. Secondary endpoints include associations with clinicopathologic variables (lesion site and depth, parametrial/rectovaginal/bowel involvement), and exploratory analyses of indices that may discriminate patients with severe pain.

Statistics will be performed with SPSS (v23). Categorical variables are summarized as n (%) and compared with χ² or Fisher's exact tests; continuous variables as mean ± SD (or median [min-max]) and compared with Student's t-test or Mann-Whitney U test as appropriate; within-group paired comparisons may use the Wilcoxon test. Two-sided p < 0.05 denotes statistical significance. Because this is a retrospective audit with predefined time frame and all-comer surgical inclusions, no formal sample size calculation is planned.

Risks/Benefits: This is minimal-risk research using archived pathology and existing clinical records; no additional procedures or changes to care are required. Results may clarify whether tissue-level neural metrics in DIE nodules reflect the patient's pain phenotype, potentially informing counseling, surgical planning (e.g., nerve-sparing strategies), and the development of response biomarkers for future prospective studies.

ELIGIBILITY:
Inclusion Criteria:Female, 18-55 years of age at time of surgery

Surgically treated for deep infiltrating endometriosis (DIE) with curative intent within the study period

Histopathologic confirmation of DIE on resected specimen (e.g., rectovaginal septum, uterosacral/cardinal ligaments, parametria, bowel, ureter, bladder, retrocervical/cervicovaginal sites)

Availability of archived FFPE tissue blocks adequate for H&E and immunohistochemistry (e.g., SOX10) to quantify nerve fiber density

Documented preoperative pain assessment (e.g., VAS 0-10 for dysmenorrhea, dyspareunia, dyschezia, dysuria, and/or chronic pelvic pain) obtained within ≤3 months prior to index surgery

Accessible clinical data in the medical record (demographics, gynecologic history, prior medical/surgical therapies) sufficient for planned analyses

IRB approval in place; inclusion under written informed consent or IRB waiver applicable to retrospective data/tissue use -

Exclusion Criteria:No surgical resection of DIE (e.g., diagnostic laparoscopy only) or no histopathologic confirmation of DIE

Insufficient biospecimen (no/poor-quality FFPE tissue for H&E/IHC)

Missing preoperative pain assessment (no VAS data within ≤3 months before index surgery)

Concomitant malignancy of the pelvis/abdominopelvic organs or malignancy treated within the past 5 years

Prior pelvic radiotherapy or major pelvic/nerve ablative surgery that precludes meaningful pain attribution

Acute pelvic infection at time of assessment or surgery (e.g., PID, tubo-ovarian abscess)

Primary pain disorders likely to confound attribution (e.g., interstitial cystitis/bladder pain syndrome, IBS with pain as dominant symptom, centrally mediated chronic pain syndromes) without adequate documentation to separate pain sources

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women
Study Population: Women aged 18-55 with surgically confirmed deep infiltrating endometriosis (DIE) treated at tertiary referral endometriosis centers during the study period. Consecutive, real-world all-comer surgical cases are included after inadequate response to medical therapy, encompassing common DIE sites (rectovaginal septum, uterosacral/cardinal ligaments, parametria, retrocervical/cervicovaginal, bowel, ureter, bladder). All participants have archived FFPE specimens suitable for histopathology/IHC and a documented preoperative pain assessment (e.g., VAS). The cohort is observational, retrospective, with no investigational intervention.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Association between nodule-level nerve fiber density and pelvic pain severity | from 01.02.2022 to june 2025
  Nerve fiber density (SOX10-positive neural profiles per high-power field on FFPE sections of DIE nodules) will be quantified and averaged per nodule. Pelvic pain severity will be extracted from patient-reported visual analogue scale (VAS, 0-10) scores for relevant domains (e.g., dysmenorrhea, dyspareunia, dyschezia, dysuria, chronic pelvic pain). The primary analysis tests the association between nerve fiber density and VAS severity (Spearman correlation and multivariable linear regression adjusting for age, lesion site/depth, and prior treatments). Higher nerve fiber density is hypothesized to correlate with higher VAS pain scores.

CONTACTS AND LOCATIONS:
Overall Officials: baris kaya, associate professor, Principal Investigator — Basaksehir Cam ve Sakura Sehir Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Basaksehir Cam Ve Sakura Sehir Hospital, Istanbul
  - Basaksehir Cam ve Sakura City Hospital, Başakşehir Mahallesi G-434 Caddesi No: 2L Başakşehir / İSTANBUL, Istanbul

IPD SHARING:
Plan to Share IPD: No
This retrospective, single-cohort study uses de-identified data from routine care and archived tissue. Individual participant data will not be shared publicly.

REFERENCES:
- [Background] Zomer MT, Kondo W, Cavalcanti TCS, Von Linsigen R, Ferreira LRG, Carranco RC, Trippia CH, Kulak J Jr. Assessment of Nerve Fiber Density and Expression of Hormonal Receptors Within Rectosigmoid Endometriosis Nodules. J Minim Invasive Gynecol. 2022 Feb;29(2):265-273. doi: 10.1016/j.jmig.2021.08.008. Epub 2021 Aug 17. PMID 34411730
- [Background] Tokushige N, Markham R, Russell P, Fraser IS. Nerve fibres in peritoneal endometriosis. Hum Reprod. 2006 Nov;21(11):3001-7. doi: 10.1093/humrep/del260. Epub 2006 Sep 1. PMID 16950827
- [Background] McKinnon B, Bersinger NA, Wotzkow C, Mueller MD. Endometriosis-associated nerve fibers, peritoneal fluid cytokine concentrations, and pain in endometriotic lesions from different locations. Fertil Steril. 2012 Feb;97(2):373-80. doi: 10.1016/j.fertnstert.2011.11.011. Epub 2011 Dec 10. PMID 22154765
- [Background] Wang G, Tokushige N, Markham R, Fraser IS. Rich innervation of deep infiltrating endometriosis. Hum Reprod. 2009 Apr;24(4):827-34. doi: 10.1093/humrep/den464. Epub 2009 Jan 16. PMID 19151028
- [Background] Yan D, Liu X, Guo SW. Neuropeptides Substance P and Calcitonin Gene Related Peptide Accelerate the Development and Fibrogenesis of Endometriosis. Sci Rep. 2019 Feb 25;9(1):2698. doi: 10.1038/s41598-019-39170-w. PMID 30804432
- [Background] Mabrouk M, Raimondo D, Arena A, Iodice R, Altieri M, Sutherland N, Salucci P, Moro E, Seracchioli R. Parametrial Endometriosis: The Occult Condition that Makes the Hard Harder. J Minim Invasive Gynecol. 2019 Jul-Aug;26(5):871-876. doi: 10.1016/j.jmig.2018.08.022. Epub 2018 Aug 31. PMID 30176361
- [Background] Koninckx PR, Meuleman C, Demeyere S, Lesaffre E, Cornillie FJ. Suggestive evidence that pelvic endometriosis is a progressive disease, whereas deeply infiltrating endometriosis is associated with pelvic pain. Fertil Steril. 1991 Apr;55(4):759-65. doi: 10.1016/s0015-0282(16)54244-7. PMID 2010001